CLINICAL TRIAL: NCT05310643
Title: Nivolumab and Ipilimumab in Patients With dMMR and/or MSI Metastatic Colorectal Cancer Resistant to Anti-PD1 Monotherapy: An Open-label Phase II GERCOR Trial (NIPIRESCUE)
Brief Title: Nivolumab and Ipilimumab in Anti-PD1-Resistant dMMR/MSI mCRC
Acronym: NIPIRESCUE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIPIRESCUE G-113
Record Dates: First submitted 2022-01-28; First posted 2022-04-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: dMMR; MSI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment phase (Experimental): Induction therapy: Nivolumab 240 mg + ipilimumab 1 mg/kg every 3 weeks for 4 dosing cycles (4 infusions of nivolumab and ipilimumab).
  Maintenance therapy: Nivolumab 480 mg every 4 weeks (21 infusions).
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Induction therapy with nivolumab 240 mg; 4 infusions, every 3 weeks.
  Maintenance therapy with nivolumab 480 mg; 21 infusions, every 4 weeks.
  Other Names: Opdivo
Drug: Ipilimumab — Induction therapy with ipilimumab 1 mg/kg; 4 infusions, every 3 weeks.
  Other Names: Yervoy

SUMMARY:
NIPIRESCUE evaluates nivolumab and ipilimumab in patients with MSI/dMMR mCRC resistant to anti-PD1 monotherapy and previously treated with fluoropyrimidine, oxaliplatine, irinotecan, and anti- vascular endothelial growth factor (VEGF) or anti- epidermal growth factor receptor (EGFR) therapy.

DETAILED DESCRIPTION:
NIPIRESCUE is a national, single-arm, open-label phase II study, evaluating nivolumab and ipilimumab in patients with MSI/dMMR mCRC resistant to anti-PD1 monotherapy and previously treated with fluoropyrimidine, oxaliplatine, irinotecan, and VEGF or anti-EGFR therapy. Patients after inclusion will receive: Induction therapy with nivolumab 240 mg and ipilimumab 1 mg/kg every 3 weeks for 4 dosing cycles (4 infusions of nivolumab and ipilimumab) and maintenance therapy with by nivolumab 480 mg every 4 weeks (21 infusions). The primary endpoint is ORR at 24 weeks (6 months) from the beginning of the treatment evaluated by RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated patient informed consent form and willingness to comply with all study procedures and availability for the study duration,
2. Age ≥ 18 years,
3. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0, 1, and 2,
4. Histologically confirmed colorectal adenocarcinoma,
5. Documented metastatic disease not suitable for complete surgical resection,
6. Disease progression per iRECIST criteria (i.e., iCPD: immune confirmed PD) during monotherapy with anti-PD1 monoclonal antibody or less than 6 months after the discontinuation of anti-PD1 monoclonal antibody
7. Disease progression during, after, or patients who are intolerant or have contraindications to approved standard therapies for the metastatic disease, which must include at least: • Fluoropyrimidine, oxaliplatin, and irinotecan, • Anti-EGFR therapy if wild-type RAS, • Anti-VEGF therapy,
8. At least one measurable lesion as assessed by CT-scan or magnetic resonance imaging (MRI) according to RECIST 1.1 and feasibility of repeated radiological assessments,
9. dMMR and/or MSI tumor status defined by: - Loss of MMR protein expression using immunohistochemistry with four (anti-MLH1, anti-MSH2, anti-MSH6, and anti-PMS2) antibodies, - and/or ≥ two unstable markers by pentaplex polymerase chain reaction (BAT-25, BAT-26, NR-21, NR-24, and NR-27), NB: In case of loss of expression of only one MMR protein immunohistochemistry, it is necessary to confirm the tumor is MSI using pentaplex PCR.

   NB: In cases with two unstable markers, comparison with matching normal tissue is required.

   NB: Agreement of the Sponsor (GERCOR) is mandatory to include the patient (the patient's file will be verified to confirm MSI/dMMR status before inclusion [an anonymized fax] and confirmation of a patient's allocation will be sent by mail to the Investigator within 24h).
10. For all patients, a new biopsy must be performed to obtain fresh anti-PD1 resistant tumor tissue prior to study treatment initiation,
11. For all patients, archival formalin-fixed paraffin-embedded tissue (FFPE) blocks and/or FFPE unstained slides (minimum of 30 positively charged slides representative of tumor tissue and non-tumor adjacent prior to anti-PD1 therapy (i.e., primary or metastatic site naïve of immunotherapy) must be submitted to the central laboratory,
12. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 7 days prior inclusion: - Adequate hematological status (White blood cell > 2000/μL; o Neutrophils > 1500/μL; Platelets > 100.000/μL; Hemoglobin > 10.0 g/dL; - Adequate renal function: Serum creatinine level < 120 μM; Clearance > 50 ml/min (Modification of the Diet in Renal Disease [MDRD] or Cockcroft and Gault, - Adequate liver function: Serum bilirubin ≤ 1.5 x upper normal limit (ULN); Alkaline phosphatase (ALP) ≤ 3.0 x ULN; Alanine aminotransferase (ALT) ≤ 3.0 x ULN; Aspartate aminotransferase (AST) ≤ 3.0 x ULN; Hemostasis: Prothrombin time (PT)/International normalized ratio (INR) and activated partial PT (aPTT) ≤ 1.5 x ULN unless participants are receiving anticoagulant therapy and their INR is stable and within the recommended range for the desired level of anticoagulation,
13. Females of childbearing potential must have negative serum pregnancy test within 7 days before starting study treatment,
14. Women of childbearing potential should use effective contraception during treatment and at least 5 months thereafter.
15. Registration in a national health care system (Protection Universelle Maladie [PUMa] included)

Exclusion Criteria:

1. Known brain metastases or leptomeningeal metastases,
2. Persistence of toxicities related to prior treatments (chemotherapies or anti-P1 therapies) grade > 1 (NCI CTCAE v 5.0; except dysthyroidism, adrenal gland deficiency, alopecia, fatigue or oxaliplatin-induced peripheral sensory neuropathy which can be ≥ grade 2),
3. Discontinuation of anti-PD1 treatment due to treatment-related adverse event (AE) grade > 2 (NCI CTCAE v 5.0),
4. Prior treatment with an anti-LAG-3, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including prior therapy with anti-tumor vaccines or other immuno-stimulatory antitumor agents, except anti-PD1 antibodies,
5. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, radiotherapy, immunotherapy),
6. Major surgical procedure within 4 weeks prior to initiation of study treatment,
7. Patients receiving any investigational drug, biological, immunological therapy within the previous 21 days before study treatment,
8. Patients with an active, known, or suspected autoimmune disease. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to be enrolled,
9. History of interstitial lung disease or pneumonitis,
10. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of inclusion.

    NB : Exceptions to this criterion: - Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease, - Systemic corticosteroids at physiologic doses not exceeding strictly 10 mg/day of prednisone or its equivalent,
11. Prior malignancy active within the previous 3 years, except for: - Locally curable cancers that have been apparently cured (e.g. squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast), - Lynch syndrome-related non-colorectal cancer in complete remission for > 1 year,
12. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test prior to randomization) virus (HBV) or hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection. Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid.
13. Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
14. Any serious or uncontrolled medical disorder that, in the opinion of Investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the participant to receive protocol therapy, or interfere with the interpretation of study results,
15. Known allergy/hypersensitivity to any component of study agents,
16. Administration of a (attenuated) live vaccine within 28 days of planned start of study therapy of known need for this vaccine during treatment,
17. Patient under a legal protection regime (guardianship, curatorship, judicial safeguard) or administrative decision or incapable of giving his/her consent,
18. Impossibility of submitting to the medical follow-up of the study for geographical, social, or psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | At week 24 (6 months)
  ORR defined as the number of patients with partial or complete response from the beginning of the treatment divided by the total of number of patients evaluable for the primary endpoint analysis.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | Up to 100 days after the last dose
  All grade and severe toxicities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Disease control rate (DCR) | At 24 week
  DCR by RECIST 1.1 is defined as the percentage of patients who achieve complete response, partial response, or stable disease after study treatment.
Duration of response | From the time of the first response observed (PR or CR) until documented tumor progression or death, assessed up to 3 years from inclusion
  Duration of response is measured from the time of the first response observed (partial or complete) until documented tumor progression or death.
Progression-free survival (PFS) | From beginning of treatment to progression or death due to any cause, whichever occurs first, assessed up to 3 years from inclusion
  PFS by RECIST 1.1 is defined as time from beginning of treatment to progression or death due to any cause, whichever occurs first. Death event will be assessed until the initiation of the subsequent anti-cancer therapy.
Overall survival (OS) | From beginning of treatment to death from any cause, assessed up to 3 years from inclusion
  OS is defined as the time between beginning of treatment and death from any cause. Survival data will be censored at the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Romain COHEN, MD, Principal Investigator — Saint Antoine Hospital
Locations (9):
- France (9):
  - CHU Jean Minjoz, Besançon
  - Institute Bergonie, Bordeaux
  - CHRU Lille, Lille
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint Antoine, Paris
  - CHU Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No